CLINICAL TRIAL: NCT06274112
Title: Personalized Neuromodulation Targeting Dysregulated Motivational Responses Underlying Social Avoidance Behavior
Brief Title: Using TMS to Understand Neural Processes of Social Motivation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Travis Evans, Assistant Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1K23MH135222 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Social Avoidant Behavior; Major Depressive Disorder; Social Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Phobia, Social

STUDY DESIGN:
Intervention Model Description: All participants will receive each dose of TMS in a counterbalanced order (AB or BA)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TMS A (Experimental): Active continuous thetaburst stimulation administered over right dorsolateral prefrontal cortex for 40 seconds (600 pulses total)
  Interventions: Device: TMS
- TMS B (Sham Comparator): Sham continuous thetaburst stimulation administered over right dorsolateral prefrontal cortex for 40 seconds (600 pulses total)
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — TMS will be administered using a Cool B-65 coil to a personalized right dlPFC region.

SUMMARY:
The purpose of this study is to use transcranial magnetic stimulation (TMS) to better understand the neural circuits associated with social motivation.

Participant includes four study visits each that range from 1.5 - 3.0 hours in duration over approximately a one month period. The first study visit involves answering survey questions, a clinical interview, and computer tasks. The second study visit involves a magnetic resonance imaging (MRI) scan, computer tasks, and a brief TMS protocol. The second and third study visits involve a full session of TMS followed by an MRI scan and computer tasks.

Adults in the Auburn/Apelika area who avoid social situations, experience symptoms of depression or social anxiety, and are between 25 years old and 50 years old are eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Major Depressive Disorder OR a diagnosis of Social Anxiety Disorder (assessed/confirmed at screening visit).
* Scoring above clinical threshold on a measure of social avoidant behavior (assessed/confirmed at screening visit).

Exclusion Criteria:

* Unstable medication regimen (i.e., changes in medication or dosage in past 3 months).
* Current or lifetime diagnosis of Bipolar Disorder.
* A diagnosis of substance use disorder within past 12 months.
* A diagnosis of psychotic-spectrum disorder such as Schizophrenia.
* Pregnancy or probable pregnancy.
* Medical illness or medical treatment that would preclude or inhibit study participation.
* Neurological disorder or prior neurosurgical procedure.
* History of seizures or head trauma.
* Metal implants or objects within body (e.g., pacemaker).

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Social motivation | Immediately post-intervention
  Motivational responses to facial expressions as measured by the Social Approach Avoidance Paradigm (SAAP; Evans, Esterman, & Britton, 2022). In the SAAP, participants self-report how much they would like to approach or avoid emotional facial expressions.
Neural circuit function | Immediately post-intervention
  Brain connectivity during motivational responses to facial expression during the Social Approach-Avoidance Paradigm (SAAP; Evans, Esterman, & Britton, 2022) and during resting state conditions. In the SAAP, participants self-report how much they would like to approach or avoid emotional facial expressions. During resting state conditions, participants simply lie still with their eyes open without completing any type of task.